CLINICAL TRIAL: NCT01739231
Title: Safety, Reactogenicity, Tolerability, Immunogenicity and Efficacy of Live Attenuated ETEC ACE527 Vaccine Administered Alone or With a Double Mutant E. Coli Heat Labile Toxin (dmLT) in Healthy Adult Volunteers
Brief Title: Live Attenuated ETEC Vaccine ACE527 With and Without dmLT Adjuvant in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAC 006
Record Dates: First submitted 2012-09-21; First posted 2012-12-03 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A of the study was masked to the participant, care provider, investigator, and outcomes assessor. Part B was open label.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACE527 alone (Experimental): In Part A of the study, subjects were split into two cohorts whereby enrollment of the second cohort depended on the safety profile of the first cohort. In Part A, subjects received three oral doses of ACE527 at 0, 1, and 2 months. For Part B of the study, eligible subjects who expressed interest of the study were administered H10407 challenge strain 5-7 months after the three-dose vaccination series.
  Interventions: Biological: ACE527; Biological: H10407 challenge strain
- ACE527 plus dmLT (Experimental): In Part A of the study, subjects were split into two cohorts whereby enrollment of the second cohort depended on the safety profile of the first cohort. In Part A, subjects received three oral doses of ACE527 with mucosal adjuvant (dmLT) at 0, 1, and 2 months. For Part B of the study, eligible subjects who expressed interest of the study were administered H10407 challenge strain 5-7 months after the three-dose vaccination series.
  Interventions: Biological: ACE527; Biological: dmLT; Biological: H10407 challenge strain
- Control: Part A and B (Active Comparator): In Part A of the study, subjects were split into two cohorts whereby enrollment of the second cohort depended on the safety profile of the first cohort. In Part A, subjects received three oral doses of CeraVacx placebo at 0, 1, and 2 months. For Part B of the study, eligible subjects who expressed interest of the study were administered H10407 challenge strain 5-7 months after the three-dose vaccination series.
  Interventions: Biological: CeraVacx placebo; Biological: H10407 challenge strain
- Control: Part B only (Active Comparator): Eligible participants were screened and administered H10407 challenge strain concurrently with other arms in Part B of the study. Their results for Part B are combined with that of the Control Arm in Part A, which received three oral doses of CeraVacx placebo.
  Interventions: Biological: H10407 challenge strain

INTERVENTIONS:
Biological: ACE527 — 3x10^9 cfu ACE527 vaccine strain. Comprised of three genetically attenuated and engineered strains of E. coli, with antigen profiles covering a wide range of ETEC surface colonization factor antigens (CFA/I, CFA/II [CS1, CS2, CS3] and CFA/IV [CS5, CS6]) and also expressing LTB, the inactive subunit of LT (ETEC heat labile toxin). The constituent strains of ACE527 were:
  * ACAM2025: a live, attenuated, CFA/I, LTB positive strain
  * ACAM2022: a live, attenuated, CS5, CS6, LTB positive strain, and
  * ACAM2027: a live, attenuated, CS1, CS2, CS3, LTB positive strain.
  Arms: ACE527 alone; ACE527 plus dmLT
Biological: dmLT — A derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine (13). These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
  Other Names: LT(R192G/L211A)
  Arms: ACE527 plus dmLT
Biological: CeraVacx placebo — CeraVacx® is used to neutralize gastric acidity upon ingestion of vaccine. It was also used as the placebo in this study. CeraVacx® was prepared from the commercial product (Cera Products, Inc.); 9.5 grams were added to sterile water for each dose and mixed. Each dose contained 7 grams of rice syrup, 2 grams of sodium bicarbonate, and 0.5 grams of trisodium citrate.
  Arms: Control: Part A and B
Biological: H10407 challenge strain — Approximately 2 x 10^7 cfu of the fully virulent ETEC strain. Previously administered to 91 volunteers at this challenge dose by the CIR clinical team over the previous 4 years in conjunction with other Phase 1/2b trials.
  Other Names: ST+, LT+, CFA/I toxin

SUMMARY:
This is a research study about an experimental (investigational) oral ETEC vaccine (ACE527). ACE527 is a live attenuated vaccine that is being made to prevent disease from enterotoxigenic Escherichia coli (ETEC), which causes watery diarrhea, largely in children living in developing countries and in travelers to those countries. This research study is also testing an investigational adjuvant called dmLT. An adjuvant is something that is added to a vaccine to make it work better. The purpose of this study is two-fold. First, Part A aims to find out if the vaccine by itself or the vaccine combined with the adjuvant is safe, tolerable, and initiates an immune response. Second, Part B aims to find out if the vaccine by itself or the vaccine combined with the adjuvant prevents diarrheal disease when challenged with ETEC H10407. About 60 healthy adults, ages 18-50, will participate in Part A, and they will be required to stay in the research facility for several nights for the first dose, but will not be required to stay overnight for the second and third doses. Participants will be assigned to receive either the vaccine alone, the vaccine with adjuvant, or placebo by mouth. Study procedures include: stool samples, blood samples, and documentation of side effects. Participants will be involved in study related procedures for about 8 months.

Interested volunteers from Part A will along with volunteers who were never vaccinated in Part A will return to participate in Part B. These volunteers will be required to stay overnight in the research facility for several nights after challenge, after which they will be treated with antibiotics and sent home. Study procedures include stool samples, blood samples, and documentation of infection with ETEC H10407. If the vaccine with/without adjuvant is effective, the volunteers should not development diarrhea, but if the vaccine with/without adjuvant is not effective, the volunteers will have diarrhea for a few days.

DETAILED DESCRIPTION:
This study is a clinical trial in healthy adult volunteers to evaluate the safety, immunogenicity and efficacy of a live attenuated ETEC vaccine, ACE527, with and without a mucosal adjuvant, dmLT. This study was designed initially as a single site, Phase 1, double-blind, randomized, placebo-controlled, clinical trial in healthy adult volunteers to evaluate the safety and immunogenicity of a live attenuated ETEC vaccine, ACE527, with and without a mucosal adjuvant, dmLT (Part A). The addition of a challenge step provides a unique opportunity to evaluate the efficacy of the new lyophilized formulation of ACE527 vaccine, given in a two or three dose regimen, with and without dmLT, against wild type ETEC strain H10407 challenge (designated as Part B: Phase 2b Open Label Challenge Study). In addition, challenging the volunteers may allow for the identification of immune correlates of protection, taking advantage of newly available technologies (immune proteomics, transcriptomics, etc.)

ACE527 comprises three genetically attenuated and engineered strains of E. coli, with antigen profiles covering a wide range of ETEC surface colonization factor antigens (CFA/I, CFA/II [CS1, CS2, CS3] and CFA/IV [CS5, CS6]) and also expressing LT-B, the inactive subunit of LT (ETEC heat labile toxin). LT(R192G/L211A), or dmLT, is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine.

Volunteers were enrolled in Part A into each of two separate Cohorts. Cohort 1 and 2 volunteers received 10^10 colony-forming units (cfu) total dose of ACE527, 10^10 cfu total dose of ACE527 with 25 µg dmLT, or placebo at 0, 1, and 2 months. Enrollment and dosing of Cohort 2 was dependent on an acceptable safety profile of the first dose of Cohort 1, based on evaluation of data up until Day 3 by the Safety Review Committee (SRC). The first immunization of each Cohort was administered in the Center for Immunization Research (CIR) Inpatient Unit, followed by 72 hours of direct post-immunization observation. The SRC met after the first dose of cohort to determine continuation of volunteer dosing on an outpatient basis, and enrollment of Cohort 2. The SRC met again after the first dose of Cohort 2 after concluding that the first dose appeared safe and well tolerated, subsequent doses would be administered on an outpatient basis. Safety was assessed by solicited symptoms/subject memory aid and laboratory evaluations. Adverse events (AE)s were graded according to standardized criteria. The immunogenicity outcome measures of interest include serum immunoglobulin G (IgG) and immunoglobulin A (IgA) antibodies by enzyme-linked immunosorbent assay (ELISA) against all vaccine antigens, cytokine assays, B and T cell memory responses, shedding profile of ACE527, and vaccine specific mucosal IgA responses.

Part B challenge cohorts were recruited among those participating in Part A; plus additional unvaccinated control volunteers sufficient to enroll up to a total of 60 recruited, as needed. Volunteers in the Phase 2b study were enrolled and challenged in 2-4 cohorts due to the CIR Inpatient Unit capacity of 30 beds. A minimum of 8-10 controls were challenged with each cohort of vaccinees to ensure comparability of attack rates across challenge cohorts. Volunteers were admitted as inpatients and challenged, with approximately 2 x 10^7 cfu of the fully virulent ETEC strain, H10407, followed by 5 days of direct observation. A Data Review Committee (DRC) will be convened to review the clinical data for all challenged volunteers and verify all outcomes per protocol definitions before any vaccine efficacy assessments were made.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy adults between 18 and 50 years of age at the time of enrollment.
2. General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of PI.
3. Negative pregnancy test at screening and before the first (V0), second (V28), and third vaccinations (V56) for female volunteers of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female volunteers unable to bear children must have this documented (e.g. tubal ligation or hysterectomy) or must have negative pregnancy tests.
4. Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
5. Completion of a training session and demonstrated comprehension of the protocol procedures and knowledge of ETEC associated illness by passing a written examination (70% pass score).
6. Availability for the study duration, including all planned follow-up visits.
7. Received at least 2 doses of ACE527 vaccine alone or in combination with 25 ug dmLT 4-6 months prior to challenge (Part B only)

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition which in the opinion of the investigator precludes participation in the study. Some medical conditions which are adequately treated and stable would not preclude entry into the study. These conditions might include stable asthma controlled with inhalers or mild hypertension stably controlled with a single agent.
2. Significant abnormalities in screening hematology, or serum chemistry as determined by PI or PI in consultation with the Medical Officer and sponsor.
3. Presence in the serum of HIV antibody, HBsAg, or HCV antibody.
4. Evidence of IgA deficiency (serum IgA < 7 mg/dl or limit of detection of assay).
5. Evidence of current excessive alcohol consumption or drug dependence.
6. Volunteers whose Body Mass Index (BMI) is less than 19.0 or greater than 34.0 (kg/m2)
7. Recent vaccination or receipt of an investigational product (within 30 days before vaccination).
8. Intention to donate blood or blood products within one month following the completion of study participation (note: The Red Cross will not allow blood donations for 1 year following participation in an investigational research study).
9. Any other criteria which, in the investigator's opinion, would compromise the ability of the volunteer to participate in the study, the safety of the study, or the results of the study
10. Working as a food handler, in child-care or as a healthcare worker with direct patient contact.
11. Have household contacts who are <2 years old or >80 years old or infirm or immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease).
12. Abnormal stool pattern (fewer than 3 per week or more than 3 per day).
13. Regular (≥ weekly) use of laxatives, antacids, or other agents to lower stomach acidity.
14. Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding the first vaccination or planned use during the active study period.
15. Symptoms consistent with Traveler's Diarrhea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within two years prior to dosing, OR planned travel to endemic countries during the length of the study.
16. Vaccination for or ingestion of ETEC, cholera, or LT toxin within 3 years prior to dosing.
17. Use of antibiotics during the 7 days before dosing or proton pump inhibitors, H2 blockers or antacids within 48hours prior to dosing.
18. History of diarrhea in the 7 days prior to vaccination (outpatient diarrhea is defined as ≥ 3 unformed (grade 3 or greater) loose stools in 24 hours).
19. Known allergy to two of the three following antibiotics: Ciprofloxacin, amoxicillin, and/or trimethoprim/sulfamethoxazole

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton D Harro, MD, ScM, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research (CIR) at Johns Hopkins School of Public Health (JHSPH), Baltimore, Maryland, United States

REFERENCES:
- [Derived] Harro C, Louis Bourgeois A, Sack D, Walker R, DeNearing B, Brubaker J, Maier N, Fix A, Dally L, Chakraborty S, Clements JD, Saunders I, Darsley MJ. Live attenuated enterotoxigenic Escherichia coli (ETEC) vaccine with dmLT adjuvant protects human volunteers against virulent experimental ETEC challenge. Vaccine. 2019 Mar 28;37(14):1978-1986. doi: 10.1016/j.vaccine.2019.02.025. Epub 2019 Feb 21. PMID 30797634

RESULTS

PARTICIPANT FLOW:
Groups:
- ACE527 Alone: In Part A, subjects received three oral doses of ACE527 at 0, 1, and 2 months. For Part B of the study, eligible subjects who expressed interest of the study were administered H10407 challenge strain 5-7 months after the three-dose vaccination series.
- ACE527 Plus dmLT: In Part A, subjects received three oral doses of ACE527 with mucosal adjuvant (dmLT) at 0, 1, and 2 months. For Part B of the study, eligible subjects who expressed interest of the study were administered H10407 challenge strain 5-7 months after the three-dose vaccination series.
- Control: Part A and B: In Part A, subjects received three oral doses of CeraVacx placebo at 0, 1, and 2 months. For Part B of the study, eligible subjects who expressed interest of the study, plus participants who had not participated in Part A, were administered H10407 challenge strain 5-7 months after the three-dose vaccination series.
- Control: Part B Only: Participants who were recruited after Part A of the study, for Part B. Participants were administered H10407 challenge strain concurrently with other subjects in Part B.
Period: Part A
Arm/Group | ACE527 Alone | ACE527 Plus dmLT | Control: Part A and B | Control: Part B Only
Started | 24 | 24 | 12 | 0
Received All 3 Vaccinations | 21 | 20 | 12 | 0
Completed | 20 | 17 | 12 | 0
Not Completed | 4 | 7 | 0 | 0
Period: Part B
Arm/Group | ACE527 Alone | ACE527 Plus dmLT | Control: Part A and B | Control: Part B Only
Started | 20 | 17 | 12 | 21
Challenged | 13 | 13 | 10 | 21
Completed | 13 | 12 | 10 | 19
Not Completed | 7 | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part A: ACE527 Alone: Participants assigned to receiving three oral doses of ACE527 only at 0, 1, and 2 months.
- Part A: ACE527 Plus dmLT: Participants assigned to receiving three oral doses of ACE527 plus mucosal adjuvant (dmLT) at 0, 1, and 2 months.
- Part A: Placebo: Participants assigned to receiving three oral doses of CeraVacx placebo at 0, 1, and 2 months.
- Part B: ACE527 Alone: Participants assigned to receiving three oral doses of ACE527 only at 0, 1, and 2 months and participated in Part B of the study.
- Part B: ACE527 Plus dmLT: Participants assigned to receiving three oral doses of ACE527 plus mucosal adjuvant (dmLT) at 0, 1, and 2 months and participated in Part B of the study.
- Part B: Control: Participants assigned to receiving three oral doses of CeraVacx placebo at 0, 1, and 2 months and participated in Part B of the study, plus additional participants who did not participate in Part A.
- Total: Total of all reporting groups
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control | Total
Number analyzed (Participants) | 24 | 24 | 12 | 13 | 13 | 31 | 117
Age, Continuous [Mean (Full Range); unit: years] — Population: 13 participants receiving ACE527 alone, 13 receiving ACE527 plus dmLT, and 12 receiving placebo participated in both Part A and Part B; and 21 participated in Part B only. Each part of the study was analyzed separately.
  years
    Part A: number analyzed (Participants) | 24 | 24 | 12 | 0 | 0 | 0 | 60
    Part A | 35.8 [21 to 48] | 37.6 [19 to 49] | 37.0 [26 to 49] |  |  |  | 36.8 [19 to 49]
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 13 | 31 | 57
    Part B |  |  |  | 37.0 [21 to 49] | 37.6 [27 to 49] | 36.5 [23 to 49] | 36.9 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 13 participants receiving ACE527 alone, 13 receiving ACE527 plus dmLT, and 12 receiving placebo participated in both Part A and Part B; and 21 participated in Part B only. Each part of the study was analyzed separately.
  Participants
    Part A: number analyzed (Participants) | 24 | 24 | 12 | 0 | 0 | 0 | 60
    Part A: Female | 7 | 9 | 1 | 0 | 0 | 0 | 17
    Part A: Male | 17 | 15 | 11 | 0 | 0 | 0 | 43
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 13 | 31 | 57
    Part B: Female | 0 | 0 | 0 | 4 | 6 | 6 | 16
    Part B: Male | 0 | 0 | 0 | 9 | 7 | 25 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 13 participants receiving ACE527 alone, 13 receiving ACE527 plus dmLT, and 12 receiving placebo participated in both Part A and Part B; and 21 participated in Part B only. Each part of the study was analyzed separately.
  Participants
    Part A: number analyzed (Participants) | 24 | 24 | 12 | 0 | 0 | 0 | 60
    Part A: Hispanic or Latino | 2 | 1 | 1 | 0 | 0 | 0 | 4
    Part A: Not Hispanic or Latino | 22 | 23 | 11 | 0 | 0 | 0 | 56
    Part A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 13 | 31 | 57
    Part B: Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 1 | 3
    Part B: Not Hispanic or Latino | 0 | 0 | 0 | 12 | 12 | 30 | 54
    Part B: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 13 participants receiving ACE527 alone, 13 receiving ACE527 plus dmLT, and 12 receiving placebo participated in both Part A and Part B; and 21 participated in Part B only. Each part of the study was analyzed separately.
  Participants
    Part A: number analyzed (Participants) | 24 | 24 | 12 | 0 | 0 | 0 | 60
    Part A: American Indian or Alaska Native | 1 | 0 | 0 |  |  |  | 1
    Part A: Asian | 0 | 0 | 0 |  |  |  | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  |  | 0
    Part A: Black or African American | 20 | 21 | 12 |  |  |  | 53
    Part A: White | 3 | 3 | 0 |  |  |  | 6
    Part A: More than one race | 0 | 0 | 0 |  |  |  | 0
    Part A: Unknown or Not Reported | 0 | 0 | 0 |  |  |  | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 13 | 31 | 57
    Part B: American Indian or Alaska Native |  |  |  | 1 | 0 | 0 | 1
    Part B: Asian |  |  |  | 0 | 0 | 0 | 0
    Part B: Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0 | 0 | 0
    Part B: Black or African American |  |  |  | 10 | 10 | 29 | 49
    Part B: White |  |  |  | 2 | 3 | 2 | 7
    Part B: More than one race |  |  |  | 0 | 0 | 0 | 0
    Part B: Unknown or Not Reported |  |  |  | 0 | 0 | 0 | 0
Height [Mean (Full Range); unit: inches] — Population: 13 participants receiving ACE527 alone, 13 receiving ACE527 plus dmLT, and 12 receiving placebo participated in both Part A and Part B; and 21 participated in Part B only. Each part of the study was analyzed separately.
  inches
    Part A: number analyzed (Participants) | 24 | 24 | 12 | 0 | 0 | 0 | 60
    Part A | 69.4 [59 to 76] | 67.4 [61 to 73] | 69.1 [65 to 73] |  |  |  | 68.5 [59 to 76]
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 13 | 31 | 57
    Part B |  |  |  | 70.0 [65 to 74] | 66.7 [61 to 75] | 69 [63 to 74] | 68.7 [61 to 75]
Weight [Mean (Full Range); unit: pounds] — Population: 13 participants receiving ACE527 alone, 13 receiving ACE527 plus dmLT, and 12 receiving placebo participated in both Part A and Part B; and 21 participated in Part B only. Each part of the study was analyzed separately.
  pounds
    Part A: number analyzed (Participants) | 24 | 24 | 12 | 0 | 0 | 0 | 60
    Part A | 190.3 [127 to 242] | 171.7 [119 to 223] | 176.2 [150 to 232] |  |  |  | 180.0 [119 to 242]
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 13 | 31 | 57
    Part B |  |  |  | 197.8 [155 to 249] | 176.5 [122 to 226] | 184.5 [141 to 247] | 185.7 [122 to 249]

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Serious Adverse Events and Adverse Events Leading to Withdrawal
Description: Unsolicited adverse events were collected throughout Part A of the study, were graded for severity, and assessed for relationship to vaccine. Withdrawal from the study due to adverse event was determined at the discretion of the study staff.
Time Frame: up to 1 month after last vaccination (3 months)
Population: Participants in Part A of the study who received at least one dose of the study product.
Measure: Number; unit: adverse events
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo
Number analyzed (Participants) | 24 | 24 | 12
adverse events
  Serious adverse event | 0 | 0 | 0
  Adverse event leading to withdrawal | 0 | 1 | 0

2. Primary Outcome: Part A: Number of Participants Experiencing Unsolicited Adverse Events, by Severity and Relationship to Vaccination
Description: Unsolicited adverse events were collected throughout Part A of the study, were graded for severity, and assessed for relationship to vaccine. Generally, mild severity is discomfort with no disruption of normal daily activities and relieved with or without symptomatic treatment; moderate severity is discomfort sufficient to reduce or affect normal daily activity somewhat and only partially relieved with symptomatic treatment; and severe is discomfort sufficient to reduce or affect normal daily activity considerably; prevents regular activities, and not relieved with symptomatic treatment. Additional description of severity for diarrhea, body temperature, and vomiting is described in the protocol.
Time Frame: up to 1 month after last vaccination (3 months)
Population: Participants in Part A of the study who received at least one dose of the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo
Number analyzed (Participants) | 24 | 24 | 12
Participants
  Not related: Mild | 10 | 9 | 4
  Not related: Moderate | 8 | 2 | 3
  Not related: Severe | 0 | 1 | 0
  Related: Mild | 2 | 6 | 0
  Related: Moderate | 0 | 2 | 1
  Related: Severe | 0 | 1 | 0

3. Primary Outcome: Part A: Number of Solicited Reactions
Description: Solicited reactions were collected 1 week after each vaccination.
Time Frame: up to 1 week after each vaccination (at 0, 1, and 2 months)
Population: Participants in Part A of the study who received at least one dose of the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo
Number analyzed (Participants) | 24 | 24 | 12
Participants
  Fever | 1 | 2 | 0
  Nausea | 4 | 3 | 0
  Vomiting | 2 | 1 | 1
  Abdominal Pain | 3 | 7 | 2
  Urgency of Defecation | 4 | 6 | 1
  Borborygmus (gurgling) | 6 | 6 | 2
  Malaise | 1 | 2 | 1
  Headache | 5 | 7 | 1
  Anorexia | 3 | 4 | 1
  Chills | 0 | 1 | 1
  Loose stools | 5 | 11 | 2
  Diarrhea | 1 | 1 | 0
  Temperature | 0 | 0 | 0
  Any reaction | 12 | 15 | 4

4. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Description: Defined as a four-fold rise or greater in geometric mean titer.
Time Frame: Vaccination 1 Day 3 and 7; Vaccination 2 pre-vaccination, Day 3, and Day 7; Vaccination 3 pre-vaccination, Day 7, and Week 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 3 | 0 | 1 | 0
  Vaccination 1: Day 7 | 0 | 7 | 12
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 2 | 0
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 3 | 0 | 2 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 22 | 22
  Vaccination 2: Day 7 | 0 | 12 | 10
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 1 | 3
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 11 | 13
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 1 | 1

5. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 3 | 0.93 [0.690 to 1.248] | 1.02 [0.828 to 1.261] | 0.83 [0.711 to 0.971]
  Vaccination 1: Day 7 | 1.04 [0.759 to 1.424] | 3.39 [1.865 to 6.152] | 5.05 [2.646 to 9.639]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.87 [0.698 to 1.084] | 1.13 [0.842 to 1.511] | 1.03 [0.829 to 1.274]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 22
  Vaccination 2: Day 3 | 0.97 [0.754 to 1.245] | 1.11 [0.858 to 1.432] | 0.94 [0.703 to 1.269]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.08 [0.767 to 1.528] | 4.14 [2.398 to 7.161] | 3.08 [2.232 to 4.237]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.97 [0.693 to 1.355] | 1.23 [0.940 to 1.602] | 1.38 [0.949 to 2.017]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.96 [0.730 to 1.272] | 4.15 [2.557 to 6.733] | 5.62 [2.953 to 10.7]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.05 [0.746 to 1.480] | 1.04 [0.766 to 1.406] | 1.05 [0.723 to 1.531]

6. Primary Outcome: Part A: Geometric Mean Titer of Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Time Frame: Pre and day 7 post all vaccinations; day 3 post-vaccination 1 and 2; week 4 post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 0.326 [0.231 to 0.460] | 0.387 [0.263 to 0.569] | 0.318 [0.226 to 0.448]
  Vaccination 1: Day 3 | 0.303 [0.203 to 0.451] | 0.395 [0.272 to 0.574] | 0.264 [0.189 to 0.369]
  Vaccination 1: Day 7 | 0.339 [0.228 to 0.504] | 1.310 [0.708 to 2.425] | 1.606 [0.837 to 3.081]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.284 [0.197 to 0.409] | 0.436 [0.298 to 0.639] | 0.334 [0.242 to 0.462]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 22
  Vaccination 2: Day 3 | 0.316 [0.208 to 0.480] | 0.457 [0.323 to 0.647] | 0.306 [0.228 to 0.411]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0.353 [0.233 to 0.535] | 1.603 [0.951 to 2.700] | 0.998 [0.675 to 1.475]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.316 [0.248 to 0.402] | 0.465 [0.333 to 0.649] | 0.437 [0.297 to 0.642]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.314 [0.214 to 0.461] | 1.573 [0.976 to 2.533] | 1.775 [1.038 to 3.036]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0.343 [0.229 to 0.513] | 0.413 [0.278 to 0.615] | 0.332 [0.240 to 0.460]

7. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Description: Defined as a four-fold rise or greater in geometric mean titer.
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 3 | 0 | 0 | 0
  Vaccination 1: Day 7 | 0 | 18 | 12
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 4 | 1
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 0 | 3 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 5 | 1
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 1 | 0
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 7 | 3
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 0 | 0

8. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 3 | 0.90 [0.807 to 0.995] | 0.95 [0.880 to 1.032] | 0.89 [0.785 to 1.013]
  Vaccination 1: Day 7 | 0.96 [0.854 to 1.080] | 10.95 [6.655 to 18.0] | 6.45 [3.598 to 11.6]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.92 [0.802 to 1.062] | 1.47 [1.121 to 1.927] | 1.06 [0.843 to 1.342]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 1.00 [0.857 to 1.164] | 1.65 [1.105 to 2.475] | 1.07 [0.856 to 1.337]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0.92 [0.828 to 1.025] | 1.99 [1.388 to 2.847] | 1.58 [1.220 to 2.048]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.93 [0.753 to 1.142] | 1.20 [0.927 to 1.544] | 1.01 [0.789 to 1.283]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.89 [0.740 to 1.071] | 2.65 [1.820 to 3.855] | 1.62 [1.142 to 2.303]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0.89 [0.740 to 1.071] | 0.96 [0.818 to 1.118] | 0.84 [0.692 to 1.023]

9. Primary Outcome: Part A: Geometric Mean Titer of Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Time Frame: Pre and day 7 post all vaccinations; day 3 post-vaccination 1 and 2; week 4 post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 0.175 [0.139 to 0.221] | 0.183 [0.152 to 0.221] | 0.178 [0.144 to 0.219]
  Vaccination 1: Day 3 | 0.157 [0.128 to 0.192] | 0.175 [0.145 to 0.210] | 0.158 [0.132 to 0.191]
  Vaccination 1: Day 7 | 0.168 [0.131 to 0.216] | 2.008 [1.235 to 3.266] | 1.146 [0.705 to 1.865]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.162 [0.133 to 0.197] | 0.269 [0.205 to 0.354] | 0.186 [0.146 to 0.236]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 0.175 [0.136 to 0.225] | 0.307 [0.207 to 0.455] | 0.179 [0.143 to 0.223]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0.161 [0.131 to 0.198] | 0.365 [0.250 to 0.532] | 0.274 [0.209 to 0.358]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.171 [0.125 to 0.233] | 0.208 [0.167 to 0.258] | 0.186 [0.146 to 0.236]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.164 [0.121 to 0.222] | 0.460 [0.320 to 0.663] | 0.299 [0.215 to 0.416]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Week 4 | 0.164 [0.121 to 0.222] | 0.173 [0.142 to 0.210] | 0.155 [0.120 to 0.201]

10. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 3 (CS3)
Description: Defined as a four-fold rise or greater in geometric mean titer.
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 3 | 0 | 1 | 1
  Vaccination 1: Day 7 | 0 | 7 | 2
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 2 | 0
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 0 | 2 | 2
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 3 | 3
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1 | 2 | 0
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 8 | 3
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Week 4 | 1 | 1 | 0

11. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 3 (CS3)
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 3 | 0.87 [0.675 to 1.133] | 1.17 [0.934 to 1.477] | 0.96 [0.707 to 1.306]
  Vaccination 1: Day 7 | 1.13 [0.961 to 1.337] | 2.95 [2.093 to 4.153] | 1.67 [1.129 to 2.473]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.89 [0.652 to 1.229] | 1.87 [1.493 to 2.333] | 1.21 [0.890 to 1.643]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 1.16 [0.864 to 1.547] | 1.66 [1.304 to 2.118] | 1.38 [0.948 to 2.019]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0.97 [0.769 to 1.214] | 2.08 [1.379 to 3.141] | 1.50 [1.102 to 2.051]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.22 [0.808 to 1.850] | 1.74 [1.343 to 2.256] | 1.40 [0.996 to 1.977]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.00 [0.679 to 1.469] | 2.68 [1.857 to 3.872] | 1.68 [1.174 to 2.402]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Week 4 | 1.14 [0.813 to 1.599] | 1.14 [0.864 to 1.497] | 0.94 [0.678 to 1.302]

12. Primary Outcome: Part A: Geometric Mean Titer of Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 3 (CS3)
Time Frame: Pre all vaccinations; day 3 post-vaccination 1 and 2; day 7 post all vaccinations; 4 weeks post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 0.292 [0.194 to 0.441] | 0.306 [0.238 to 0.395] | 0.322 [0.235 to 0.441]
  Vaccination 1: Day 3 | 0.256 [0.172 to 0.380] | 0.360 [0.250 to 0.518] | 0.310 [0.232 to 0.414]
  Vaccination 1: Day 7 | 0.331 [0.222 to 0.495] | 0.904 [0.673 to 1.214] | 0.539 [0.387 to 0.749]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.262 [0.191 to 0.359] | 0.572 [0.414 to 0.790] | 0.389 [0.314 to 0.480]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 0.338 [0.211 to 0.541] | 0.531 [0.382 to 0.740] | 0.418 [0.306 to 0.570]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0.283 [0.210 to 0.381] | 0.638 [0.403 to 1.009] | 0.466 [0.358 to 0.607]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.357 [0.236 to 0.542] | 0.509 [0.384 to 0.674] | 0.431 [0.318 to 0.584]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.292 [0.189 to 0.450] | 0.784 [0.528 to 1.164] | 0.515 [0.372 to 0.714]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0.333 [0.206 to 0.540] | 0.358 [0.266 to 0.481] | 0.288 [0.223 to 0.374]

13. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 6 (CS6)
Description: Defined as a four-fold rise or greater in geometric mean titer.
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 3 | 0 | 0 | 0
  Vaccination 1: Day 7 | 0 | 0 | 0
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 0 | 0
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 0 | 0 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 0 | 0
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 0 | 0
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 0 | 0
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Week 4 | 0 | 0 | 0

14. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 6 (CS6)
Time Frame: as for outcome 4
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 3 | 1 [1 to 1] | 0.95 [0.889 to 1.010] | 1.00 [0.987 to 1.008]
  Vaccination 1: Day 7 | 1 [1 to 1] | 0.96 [0.900 to 1.015] | 1.00 [0.987 to 1.008]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 1 [1 to 1] | 0.96 [0.900 to 1.015] | 1.00 [0.987 to 1.008]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 1 [1 to 1] | 0.97 [0.902 to 1.045] | 1.03 [0.985 to 1.086]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1 [1 to 1] | 0.96 [0.898 to 1.030] | 1.00 [0.990 to 1.003]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1 [1 to 1] | 0.97 [0.871 to 1.084] | 1.04 [0.979 to 1.110]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1 [1 to 1] | 0.96 [0.882 to 1.037] | 1.03 [0.986 to 1.078]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.01 [0.993 to 1.019] | 0.96 [0.890 to 1.030] | 1.00 [0.990 to 1.004]

15. Primary Outcome: Part A: Geometric Mean Titer of Antibody in Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 6 (CS6)
Time Frame: Pre and day 7 post all vaccinations; day 3 post-vaccination 1 and 2; week 4 post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 0.14 [0.14 to 0.14] | 0.148 [0.139 to 0.158] | 0.141 [0.140 to 0.142]
  Vaccination 1: Day 3 | 0.14 [0.14 to 0.14] | 0.140 [0.140 to 0.141] | 0.140 [0.140 to 0.141]
  Vaccination 1: Day 7 | 0.14 [0.14 to 0.14] | 0.142 [0.140 to 0.143] | 0.140 [0.140 to 0.141]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.14 [0.14 to 0.14] | 0.143 [0.138 to 0.147] | 0.14 [0.14 to 0.14]
  Vaccination 2: Day 3: number analyzed (Participants) | 12 | 22 | 21
  Vaccination 2: Day 3 | 0.14 [0.14 to 0.14] | 0.142 [0.138 to 0.147] | 0.145 [0.138 to 0.152]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0.14 [0.14 to 0.14] | 0.143 [0.138 to 0.147] | 0.14 [0.14 to 0.14]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.14 [0.14 to 0.14] | 0.145 [0.135 to 0.157] | 0.146 [0.137 to 0.156]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.14 [0.14 to 0.14] | 0.143 [0.138 to 0.148] | 0.145 [0.138 to 0.152]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Week 4 | 0.141 [0.139 to 0.143] | 0.142 [0.138 to 0.147] | 0.14 [0.14 to 0.14]

16. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 0 | 1
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 1 | 2
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 4 | 8
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 1 | 1
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 1 | 5
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 1 | 3

17. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.96 [0.881 to 1.045] | 0.97 [0.889 to 1.069] | 1.03 [0.840 to 1.255]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 1.05 [0.929 to 1.179] | 1.12 [0.985 to 1.281] | 1.24 [0.983 to 1.559]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.22 [1.076 to 1.376] | 1.68 [1.361 to 2.071] | 2.00 [1.498 to 2.677]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.92 [0.828 to 1.028] | 1.08 [0.936 to 1.243] | 1.25 [1.004 to 1.561]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.00 [0.888 to 1.117] | 1.22 [1.017 to 1.474] | 1.95 [1.396 to 2.721]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Week 4 | 1.09 [0.968 to 1.220] | 1.21 [1.062 to 1.369] | 1.56 [1.245 to 1.951]

18. Primary Outcome: Part A: Geometric Mean Titer of Antibody in Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 266 [124 to 569] | 385 [241 to 614] | 298 [191 to 466]
  Vaccination 1: Day 7 | 255 [123 to 528] | 375 [239 to 589] | 306 [197 to 476]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 278 [133 to 580] | 432 [284 to 657] | 365 [228 to 585]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 323 [148 to 707] | 646 [443 to 942] | 582 [375 to 904]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 245 [122 to 492] | 403 [245 to 663] | 350 [223 to 549]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 265 [131 to 533] | 458 [289 to 725] | 545 [336 to 884]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 289 [139 to 597] | 449 [288 to 698] | 436 [288 to 659]

19. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin A (IgA) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 11 | 9
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 2 | 4
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 6 | 6
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 1 | 4
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 3 | 3
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 1 | 4

20. Primary Outcome: Part A: Geometric Mean Fold Change in Serum ELISA Immunoglobulin A (IgA) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.99 [0.917 to 1.073] | 2.49 [1.738 to 3.574] | 2.42 [1.519 to 3.848]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 1.00 [0.900 to 1.115] | 1.44 [1.183 to 1.743] | 1.62 [1.085 to 2.435]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.00 [0.900 to 1.115] | 1.44 [1.183 to 1.743] | 1.62 [1.085 to 2.435]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.09 [1.035 to 1.153] | 1.60 [1.206 to 2.122] | 1.49 [1.045 to 2.123]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.09 [1.035 to 1.153] | 1.60 [1.206 to 2.122] | 1.49 [1.045 to 2.123]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.05 [0.937 to 1.172] | 1.23 [1.024 to 1.471] | 1.36 [0.905 to 2.037]

21. Primary Outcome: Part A: Geometric Mean Titer of Serum ELISA Immunoglobulin A (IgA) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 96.9 [34.5 to 273] | 101 [74.2 to 137] | 109 [64.7 to 184]
  Vaccination 1: Day 7 | 96.1 [33.4 to 277] | 251 [171 to 369] | 264 [163 to 428]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 97.1 [32.8 to 287] | 145 [104 to 201] | 171 [102 to 286]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 97.0 [33.8 to 279] | 189 [136 to 262] | 212 [128 to 350]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 106 [34.7 to 323] | 142 [101 to 201] | 172 [98.7 to 299]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 106 [37.7 to 297] | 163 [109 to 242] | 157 [91.7 to 268]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 102 [35.9 to 287] | 120 [88.1 to 164] | 143 [79.3 to 258]

22. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 3 (CS3)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 0 | 0
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 0 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 0 | 1
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 0 | 1
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1 | 1 | 1
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 0 | 1

23. Primary Outcome: Part A: Geometric Mean Fold Change in Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 3 (CS3)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.94 [0.888 to 0.986] | 1.02 [0.924 to 1.123] | 1.00 [0.904 to 1.112]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.97 [0.841 to 1.119] | 1.08 [0.950 to 1.228] | 1.06 [0.911 to 1.245]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.13 [0.993 to 1.295] | 1.23 [1.091 to 1.392] | 1.17 [1.009 to 1.366]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.10 [0.949 to 1.278] | 0.99 [0.921 to 1.063] | 1.04 [0.885 to 1.231]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.15 [0.896 to 1.474] | 1.00 [0.877 to 1.129] | 1.09 [0.930 to 1.267]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.11 [0.913 to 1.355] | 1.06 [0.973 to 1.156] | 1.12 [0.989 to 1.274]

24. Primary Outcome: Part A: Geometric Mean Titer of Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 3 (CS3)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 309 [117 to 815] | 341 [243 to 480] | 324 [214 to 491]
  Vaccination 1: Day 7 | 289 [112 to 742] | 347 [250 to 483] | 325 [226 to 466]
  Vaccination 2: Pre-vaccination | 299 [123 to 732] | 368 [272 to 499] | 350 [237 to 517]
  Vaccination 2: Day 7 | 350 [137 to 896] | 420 [304 to 581] | 386 [257 to 577340]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 340 [135 to 854] | 347 [239 to 504] | 324 [209 to 503]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 355 [147 to 855] | 350 [238 to 513] | 337 [213 to 533]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 344 [141 to 837] | 377 [269 to 527] | 348 [220 to 553]

25. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 6 (CS6)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 1 | 0
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 0 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 1 | 2
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 1 | 2
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 2 | 1
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 2 | 0

26. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 6 (CS6)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.96 [0.897 to 1.028] | 1.15 [1.006 to 1.316] | 0.99 [0.886 to 1.114]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.95 [0.822 to 1.102] | 1.14 [0.990 to 1.318] | 0.95 [0.845 to 1.065]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.13 [0.987 to 1.288] | 1.17 [1.024 to 1.340] | 1.15 [0.952 to 1.379]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.19 [0.967 to 1.468] | 1.26 [1.071 to 1.481] | 1.30 [1.043 to 1.614]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.27 [1.055 to 1.539] | 1.16 [0.951 to 1.421] | 1.24 [1.006 to 1.524]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.20 [1.000 to 1.433] | 1.12 [0.950 to 1.316] | 1.05 [0.886 to 1.234]

27. Primary Outcome: Part A: Geometric Mean Titer of Serum ELISA Immunoglobulin A (IgA) Response to E. Coli Surface Antigen 6 (CS6)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 15.9 [7.822 to 32.3] | 20.0 [12.3 to 32.4] | 16.3 [10.6 to 25.1]
  Vaccination 1: Day 7 | 15.3 [7.310 to 31.9] | 23.0 [14.9 to 35.4] | 16.2 [10.7 to 24.7]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 15.1 [7.659 to 29.9] | 22.8 [14.8 to 35.1] | 14.9 [9.867 to 22.4]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 17.9 [9.219 to 34.8] | 23.4 [14.8 to 37.1] | 17.1 [10.9 to 26.8]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 18.9 [9.873 to 36.3] | 23.0 [14.6 to 36.1] | 19.0 [11.8 to 30.6]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 20.2 [10.8 to 38.0] | 21.2 [13.8 to 32.5] | 18.1 [11.4 to 28.9]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 19.0 [9.965 to 36.3] | 22.2 [14.4 to 34.2] | 15.3 [9.576 to 24.5]

28. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 2 | 5
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 3 | 8
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 12 | 14
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 8 | 14
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 10 | 15
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 14 | 17

29. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.78 [0.680 to 0.883] | 1.05 [0.867 to 1.281] | 1.38 [0.986 to 1.944]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.86 [0.757 to 0.967] | 1.42 [1.126 to 1.786] | 2.04 [1.326 to 3.148]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.26 [1.117 to 1.411] | 2.51 [1.970 to 3.198] | 3.82 [2.571 to 5.674]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0.85 [0.717 to 0.997] | 2.05 [1.521 to 2.766] | 3.61 [2.281 to 5.717]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0.91 [0.783 to 1.057] | 2.38 [1.720 to 3.291] | 4.69 [3.036 to 7.258]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0.95 [0.778 to 1.165] | 3.22 [2.216 to 4.678] | 5.07 [3.354 to 7.650]

30. Primary Outcome: Part A: Geometric Mean Titer of Antibody in Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Heat Labile Toxin B Subunit (LTB)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 2469 [1707 to 3570] | 1990 [1459 to 2715] | 1903 [1456 to 2489]
  Vaccination 1: Day 7 | 1914 [1347 to 2720] | 2098 [1498 to 2938] | 2635 [1768 to 3926]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 2112 [1469 to 3036] | 2822 [2005 to 3972] | 3616 [2386 to 5479]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 3099 [2077 to 4622] | 4996 [3666 to 6808] | 6429 [4459 to 9270]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 2087 [1377 to 3163] | 4205 [2794 to 6329] | 6030 [3861 to 9419]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 2246 [1498 to 3367] | 4877 [3159 to 7531] | 7839 [5185 to 11850]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 2350 [1499 to 3683] | 6267 [4283 to 9171] | 8458 [5780 to 12375]

31. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin G (IgG) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 2 | 2
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 2 | 3
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 2 | 4
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1 | 2 | 3
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1 | 1 | 4
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1 | 1 | 3

32. Primary Outcome: Part A: Geometric Mean Fold Change in Serum ELISA Immunoglobulin G (IgG) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 1.06 [1.005 to 1.108] | 1.17 [0.982 to 1.391] | 1.22 [0.965 to 1.533]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 1.15 [0.979 to 1.348] | 1.15 [0.923 to 1.427] | 1.31 [1.021 to 1.675]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.13 [0.995 to 1.276] | 1.37 [1.119 to 1.669] | 1.68 [1.326 to 2.132]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.33 [1.049 to 1.686] | 1.41 [1.159 to 1.719] | 1.59 [1.296 to 1.947]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.30 [1.044 to 1.620] | 1.19 [0.972 to 1.462] | 1.62 [1.286 to 2.051]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.15 [0.883 to 1.502] | 1.16 [0.981 to 1.383] | 1.21 [0.967 to 1.508]

33. Primary Outcome: Part A: Geometric Mean Titer of Serum ELISA Immunoglobulin G (IgG) Response to Enterotoxigenic Escherichia Coli (ETEC) Colonization Factor 1 (CFA/I)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 633 [380 to 1055] | 748 [539 to 1037] | 646 [454 to 919]
  Vaccination 1: Day 7 | 668 [395 to 1131] | 874 [629 to 1215] | 785 [538 to 1147]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 727 [416 to 1270] | 858 [619 to 1190] | 856 [606 to 1210]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 713 [411 to 1237] | 1022 [727 to 1436] | 1116 [765 to 1630]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 842 [484 to 1465] | 1159 [794 to 1691] | 1079 [754 to 1543]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 823 [476 to 1425] | 979 [654 to 1467] | 1103 [750 to 1622]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 729 [394 to 1350] | 885 [628 to 1247] | 820 [561 to 1200]

34. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Surface Antigen 3 (CS3)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 0 | 0
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 0 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 0 | 0 | 0
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 0 | 0 | 0
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 0 | 0 | 0
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0 | 0 | 0

35. Primary Outcome: Part A: Geometric Mean Fold Change in Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Surface Antigen 3 (CS3)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.96 [0.841 to 1.094] | 0.94 [0.872 to 1.011] | 0.84 [0.753 to 0.940]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.99 [0.815 to 1.206] | 0.96 [0.878 to 1.039] | 0.90 [0.802 to 1.006]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.19 [1.066 to 1.328] | 1.14 [1.049 to 1.234] | 1.00 [0.923 to 1.086]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.01 [0.846 to 1.206] | 0.97 [0.901 to 1.049] | 0.84 [0.751 to 0.934]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.04 [0.898 to 1.203] | 0.94 [0.874 to 1.019] | 0.88 [0.776 to 1.000]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 0.97 [0.828 to 1.137] | 0.95 [0.873 to 1.038] | 0.89 [0.764 to 1.041]

36. Primary Outcome: Part A: Geometric Mean Titer of Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Surface Antigen 3 (CS3)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 1610 [1061 to 2442] | 1265 [955 to 1677] | 1809 [1262 to 2592]
  Vaccination 1: Day 7 | 1544 [972 to 2452] | 1188 [893 to 1581] | 1522 [1109 to 2088]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 1597 [958 to 2662] | 1208 [901 to 1620] | 1712 [1218 to 2408]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1915 [1203 to 3050] | 1439 [1064 to 1946] | 1939 [1349 to 2787]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1627 [1063 to 2490] | 1317 [975 to 1780] | 1648 [1140 to 2382]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1673 [1113 to 2515] | 1278 [953 to 1713] | 1733 [1173 to 2562]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1563 [992 to 2462] | 1236 [936 to 1630] | 1754 [1191 to 2584]

37. Primary Outcome: Part A: Number and Percentage of Subjects With Positive Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Surface Antigen 6 (CS6)
Description: Defined as a 2.5-fold rise or greater in geometric mean titer.
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
Participants
  Vaccination 1: Day 7 | 0 | 0 | 2
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0 | 1 | 3
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1 | 9 | 5
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 3 | 6 | 10
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 2 | 7 | 5
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 2 | 6 | 5

38. Primary Outcome: Part A: Geometric Mean Fold Change in Antibody in Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Surface Antigen 6 (CS6)
Time Frame: Day 7 post-all vaccinations; pre-vaccination 2 and 3; week 4 post-vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
fold change
  Vaccination 1: Day 7 | 0.80 [0.626 to 1.025] | 0.96 [0.785 to 1.165] | 1.00 [0.789 to 1.257]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 0.76 [0.567 to 1.012] | 1.10 [0.898 to 1.352] | 1.01 [0.704 to 1.457]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 1.38 [1.125 to 1.695] | 1.65 [1.232 to 2.205] | 1.58 [1.156 to 2.169]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 1.57 [1.161 to 2.119] | 1.49 [1.132 to 1.967] | 2.20 [1.293 to 3.745]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 1.45 [1.146 to 1.830] | 1.58 [1.220 to 2.045] | 1.77 [1.080 to 2.902]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 1.38 [1.011 to 1.874] | 1.57 [1.164 to 2.108] | 1.61 [1.073 to 2.417]

39. Primary Outcome: Part A: Geometric Mean Titer of Serum ELISA Immunoglobulin G (IgG) Response to E. Coli Surface Antigen 6 (CS6)
Time Frame: Pre and day 7 post all vaccinations; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: Placebo | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT
Number analyzed (Participants) | 12 | 24 | 24
titer
  Pre-Vaccination 1 | 36.2 [20.5 to 63.9] | 68.2 [40.1 to 116] | 54.3 [34.4 to 85.7]
  Vaccination 1: Day 7 | 29.0 [16.0 to 52.7] | 65.2 [35.2 to 121] | 54.1 [31.7 to 92.1]
  Vaccination 2: Pre-vaccination: number analyzed (Participants) | 12 | 24 | 23
  Vaccination 2: Pre-vaccination | 27.4 [14.2 to 52.9] | 75.1 [42.2 to 134] | 52.9 [30.6 to 91.6]
  Vaccination 2: Day 7: number analyzed (Participants) | 12 | 24 | 22
  Vaccination 2: Day 7 | 50.0 [26.5 to 94.4] | 112 [69.0 to 183] | 85.7 [54.2 to 136]
  Vaccination 3: Pre-vaccination: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Pre-vaccination | 56.8 [26.9 to 120] | 115 [68 to 195] | 118 [72.0 to 194]
  Vaccination 3: Day 7: number analyzed (Participants) | 12 | 21 | 21
  Vaccination 3: Day 7 | 52.5 [27.8 to 98.9] | 122 [70.2 to 212] | 95.2 [51.4 to 176]
  Vaccination 3: Week 4: number analyzed (Participants) | 12 | 23 | 21
  Vaccination 3: Week 4 | 49.9 [29.4 to 84.7] | 113 [68.4 to 185] | 86.6 [50.8 to 148]

40. Primary Outcome: Part B: Number and Percentage of Subjects Experiencing Severe Diarrhea Following H10407 Challenge Strain
Description: Severe diarrhea was defined as >800 grams of grade 3-5 stools passed over the 120-hour observation period. For episodes starting at or before 120 hours post-challenge, volunteers were followed to resolution and the total stool output weight was considered in determining whether a specific volunteer met the primary definition of severe diarrhea. The end of a diarrheal episode occurred when a volunteer did not pass any grade 3-5 stool in a 24-hour period.
  Grades were defined as follows:
  Grade 1: firm, formed (normal) Grade 2: soft, formed (normal) Grade 3: viscous opaque liquid or semi-liquid which assumes the shape of the container Grade 4: watery, non-viscous, opaque liquid which assumes the shape of the container Grade 5: clear or translucent, watery or mucoid liquid which assumes the shape of the container
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Part B: ACE527 Alone: Participants assigned to receiving three oral doses of ACE527 only at 0, 1, and 2 months and participated in Part B of the study (received fully virulent H10407 strain 5-7 months after the three-dose vaccination series).
- Part B: ACE527 Plus dmLT: Participants assigned to receiving three oral doses of ACE527 plus mucosal adjuvant (dmLT) at 0, 1, and 2 months and participated in Part B of the study (received fully virulent H10407 strain 5-7 months after the three-dose vaccination series).
- Part B: Control: Participants assigned to receiving three oral doses of CeraVacx placebo at 0, 1, and 2 months and participated in Part B of the study (received fully virulent H10407 strain 5-7 months after the three-dose vaccination series), plus additional participants who did not participate in Part A.
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
Participants
  Not severe | 6 | 10 | 10
  Severe | 7 | 3 | 21

41. Secondary Outcome: Part A: Number of Participants Shedding E. Coli on Qualification Plate
Time Frame: Pre- and day 7 post-all vaccinations; and Day 3 post-vaccinations 1 and 2; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo
Number analyzed (Participants) | 24 | 24 | 12
Participants
  Vaccination 1: Day 0 | 21 | 23 | 10
  Vaccination 1: Day 3 | 24 | 23 | 10
  Vaccination 1: Day 7 | 24 | 23 | 10
  Vaccination 2: Day 0: number analyzed (Participants) | 24 | 23 | 12
  Vaccination 2: Day 0 | 22 | 21 | 11
  Vaccination 2: Day 3: number analyzed (Participants) | 21 | 21 | 12
  Vaccination 2: Day 3 | 21 | 20 | 9
  Vaccination 2: Day 7: number analyzed (Participants) | 22 | 22 | 12
  Vaccination 2: Day 7 | 21 | 21 | 9
  Vaccination 3: Day 0: number analyzed (Participants) | 21 | 21 | 12
  Vaccination 3: Day 0 | 17 | 20 | 10
  Vaccination 3: Day 7: number analyzed (Participants) | 21 | 21 | 12
  Vaccination 3: Day 7 | 18 | 21 | 10
  Vaccination 3: Day 28: number analyzed (Participants) | 23 | 21 | 12
  Vaccination 3: Day 28 | 20 | 20 | 11

42. Secondary Outcome: Part A: Number of Participants With Positive Shedding Results for ACE527
Time Frame: Pre- and day 7 post-all vaccinations; and Day 3 post-vaccinations 1 and 2; and 4 weeks post vaccination 3
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo
Number analyzed (Participants) | 24 | 24 | 12
Participants
  Vaccination 1: Day 0 | 0 | 0 | 0
  Vaccination 1: Day 3 | 22 | 16 | 0
  Vaccination 1: Day 7 | 11 | 3 | 1
  Vaccination 2: Day 0: number analyzed (Participants) | 24 | 23 | 12
  Vaccination 2: Day 0 | 1 | 0 | 0
  Vaccination 2: Day 3: number analyzed (Participants) | 21 | 21 | 12
  Vaccination 2: Day 3 | 14 | 12 | 0
  Vaccination 2: Day 7: number analyzed (Participants) | 22 | 22 | 12
  Vaccination 2: Day 7 | 5 | 3 | 0
  Vaccination 3: Day 0: number analyzed (Participants) | 21 | 21 | 12
  Vaccination 3: Day 0 | 0 | 0 | 0
  Vaccination 3: Day 7: number analyzed (Participants) | 21 | 21 | 12
  Vaccination 3: Day 7 | 3 | 4 | 0
  Vaccination 3: Day 28: number analyzed (Participants) | 23 | 21 | 12
  Vaccination 3: Day 28 | 1 | 0 | 0

43. Secondary Outcome: Number of Participants Shedding Vaccine Strains Included in ACE527
Time Frame: 3 days after the first and second vaccinations
Population: Subjects who received the vaccination and had valid test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo
Number analyzed (Participants) | 24 | 24 | 12
Participants
  ACAM2022 strain: Vaccination 1 | 9 | 11 | 0
  ACAM2022 strain: Vaccination 2 | 4 | 7 | 0
  ACAM2025 strain: Vaccination 1: number analyzed (Participants) | 21 | 24 | 12
  ACAM2025 strain: Vaccination 1 | 6 | 5 | 0
  ACAM2025 strain: Vaccination 2: number analyzed (Participants) | 21 | 24 | 12
  ACAM2025 strain: Vaccination 2 | 5 | 7 | 0
  ACAM2027 strain: Vaccination 1 | 17 | 13 | 0
  ACAM2027 strain: Vaccination 2 | 12 | 11 | 0

44. Secondary Outcome: Part B: Number and Percentage of Subjects Experiencing Diarrhea of Any Severity
Description: Defined as mild, moderate, or severe diarrhea, specifically:
  * Mild diarrhea: 2 or 3grade 3-5 stools totaling 200 g - 400 g, or 1 grade 3-5 stool of >300 g
  * Moderate diarrhea: 4-5 grade 3-5 stools totaling >200 g or 401 - 800g
  * Severe diarrhea: > 800g grade 3-5 stool(s)
  Grades were defined as follows:
  Grade 1: firm, formed (normal) Grade 2: soft, formed (normal) Grade 3: viscous opaque liquid or semi-liquid which assumes the shape of the container Grade 4: watery, non-viscous, opaque liquid which assumes the shape of the container Grade 5: clear or translucent, watery or mucoid liquid which assumes the shape of the container
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
Participants
  None | 3 | 9 | 8
  Mild | 2 | 0 | 2
  Moderate | 1 | 1 | 0
  Severe | 7 | 3 | 21

45. Secondary Outcome: Part B: Mean Total Weight of Grade 3-5 Stools Passed Per Volunteer
Description: Grades were defined as follows:
  Grade 1: firm, formed (normal) Grade 2: soft, formed (normal) Grade 3: viscous opaque liquid or semi-liquid which assumes the shape of the container Grade 4: watery, non-viscous, opaque liquid which assumes the shape of the container Grade 5: clear or translucent, watery or mucoid liquid which assumes the shape of the container
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
grams | 1655.1 (1743.1) | 748.8 (1574.6) | 1878.2 (1729.4)

46. Secondary Outcome: Part B: Median Total Weight of Grade 3-5 Stools Passed Per Volunteer
Description: as for outcome 45
Time Frame: 5 days
Measure: Mean (Inter-Quartile Range); unit: grams
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
grams | 859 [522 to 3224] | 30 [0 to 858] | 1400 [547 to 2713]

47. Secondary Outcome: Part B: Mean Number of Grade 3-5 Stools Passed Per Volunteer
Description: as for outcome 45
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: stools
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
stools | 11.7 (9.61) | 6.0 (9.68) | 10.8 (7.99)

48. Secondary Outcome: Part B: Median Number of Grade 3-5 Stools Passed Per Volunteer
Description: as for outcome 45
Time Frame: 5 days
Measure: Median (Inter-Quartile Range); unit: stools
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
stools | 14 [0 to 27] | 1 [0 to 11] | 12 [3 to 16]

49. Secondary Outcome: Part B: Number of Subjects Experiencing Solicited Reactions Graded as Moderate or Severe
Description: Solicited reactions were generally graded as mild if there was discomfort, but no disruption of normal daily activities; moderate if if discomfort was sufficient to affect normal daily activity and partially relieved with symptomatic treatment; severe if discomfort was sufficient to affect normal daily activity considerably, prevent regular activity, and not relieved with symptomatic treatment.
Time Frame: 1 week
Population: Participants in Part A of the study who received at least one dose of the study product.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Placebo: Participants assigned to receiving three oral doses of CeraVacx placebo at 0, 1, and 2 months and participated in Part B of the study (received fully virulent H10407 strain 5-7 months after the three-dose vaccination series), plus additional participants who did not participate in Part A.
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Placebo
Number analyzed (Participants) | 13 | 13 | 31
Participants
  Nausea | 3 | 2 | 9
  Vomiting | 1 | 0 | 2
  Abdominal Pain | 0 | 4 | 13
  Urgency of Defecation | 1 | 2 | 13
  Borborygmus (gurgling) | 2 | 3 | 15
  Malaise | 3 | 3 | 11
  Headache | 2 | 2 | 5
  Anorexia | 4 | 2 | 14
  Myalgia | 0 | 1 | 6
  Chills | 2 | 2 | 8
  Temperature | 2 | 1 | 3
  Any reaction | 8 | 8 | 18

50. Secondary Outcome: Part B: Number and Percentage of Subjects Who Would Have Reduced Daily Activity
Description: When asking about adverse events, subjects were asked whether their illness resulting from ETEC would have reduced their daily activity because of their illness if they had been vacationing or traveling on business.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
Participants
  Changed planned activities: No | 9 | 8 | 10
  Changed planned activities: Yes | 4 | 5 | 21
  Stayed in bed: No | 9 | 10 | 14
  Stayed in bed: Yes | 4 | 3 | 17
  Either of the above: No | 7 | 8 | 10
  Either of the above: Yes | 6 | 5 | 21

51. Secondary Outcome: Part B: Mean Time to Onset of Diarrhea Among Subjects Who Had Diarrhea
Description: as for outcome 44
Time Frame: 5 days
Population: Among subjects who met the protocol definition of diarrhea over the observation period
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 10 | 4 | 23
hours | 51.5 (26.88) | 59.9 (27.12) | 46.4 (20.35)

52. Secondary Outcome: Part B: Quantity of H10407 Per Gram of Stool on Day 2 Post-challenge
Time Frame: 2 days after vaccination
Measure: Mean (Standard Deviation); unit: colony forming units
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 12 | 12 | 29
colony forming units | 261.30 (391.5) | 94.345 (199.1) | 154.84 (321.4)

53. Secondary Outcome: Part B: Number of Subjects Requiring Early Antibiotic Treatment and Intravenous (IV) Fluids
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
Number analyzed (Participants) | 13 | 13 | 31
Participants
  Early antibiotic treatment: No | 7 | 11 | 13
  Early antibiotic treatment: Yes | 6 | 2 | 18
  IV fluids: No | 9 | 9 | 16
  IV fluids: Yes | 4 | 4 | 15

ADVERSE EVENTS:
Time Frame: 1 month after each vaccination in Part A (total of three months); 1 month after challenge dose in Part B.
Arm/Group | Part A: ACE527 Alone | Part A: ACE527 Plus dmLT | Part A: Placebo | Part B: ACE527 Alone | Part B: ACE527 Plus dmLT | Part B: Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/12 | 0/13 | 0/13 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/12 | 1/12 | 0/12 | 0/31
Other Adverse Events (participants affected / at risk) | 18/24 | 14/24 | 7/12 | 8/13 | 9/13 | 19/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ACE527 Alone (N=24) | Part A: ACE527 Plus dmLT (N=24) | Part A: Placebo (N=12) | Part B: ACE527 Alone (N=12) | Part B: ACE527 Plus dmLT (N=12) | Part B: Control (N=31)
Fractured Right Wrist (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ACE527 Alone (N=24) | Part A: ACE527 Plus dmLT (N=24) | Part A: Placebo (N=12) | Part B: ACE527 Alone (N=13) | Part B: ACE527 Plus dmLT (N=13) | Part B: Control (N=31)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 3 | 5
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 5 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 8 | 0 | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1 | 4
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Allergy to metals (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 3 | 1 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 7
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days